CLINICAL TRIAL: NCT02353988
Title: Bicalutamide in Treating Patients With AR-positive Metastatic Triple Negative Breast Cancer
Brief Title: AR-inhibitor Bicalutamide in Treating Patients With TNBC
Acronym: Arbre
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Jinling Hospital, China (Other)
Collaborators: Wenzhou Medical University (Other); The First People's Hospital of Lianyungang (Other); Wuxi People's Hospital (Other); Nanning Second People's Hospital (Other); Jiangsu Province Hospital of Traditional Chinese Medicine (Other); The Second Hospital of Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Xiaoxiang Guan, Bicalutamide in Treating Patients With AR-positive Metastatic Triple Negative Breast Cancer, Jinling Hospital, China
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: JinlingH-001
Record Dates: First submitted 2015-01-26; First posted 2015-02-03 (Estimated); Last update posted 2015-02-03 (Estimated); Status verified 2015-01

CONDITIONS: Breast Neoplasms
Keywords: AR-positive; Androgen Antagonists; Bicalutamide; TNBC; metastatic
MeSH Terms: conditions — Breast Neoplasms; Neoplasm Metastasis | interventions — bicalutamide; Immunohistochemistry

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- bicalutamide (Experimental): This is a multi-center, open-label, phase II study to evaluate the anti-tumor activity and safety of bicalutamide administered orally daily to patients with estrogen receptor (ER)-negative/ progesterone receptor (PgR)-negative/ androgen receptor (AR)-positive metastatic breast cancer. Eligible patients will receive bicalutamide at a dose of 150mg PO daily.
  Interventions: Drug: Bicalutamide
- Physician's Choice (Active Comparator): Treatment of the Physician's Choice defined as any single agent chemotherapy, hormonal treatment or biological therapy approved for the treatment of cancer; or palliative treatment or radiotherapy, administered according to local practice, if applicable
  Interventions: Other: Physician's Choice

INTERVENTIONS:
Drug: Bicalutamide — Patients in experimental group are designated to take bicalutamide orally, 150mg on a continuous schedule. The investigator should pay attention to the patients' adverse event. Every month, the patients will be evaluated for the adverse event by the criterion National Cancer Institute Common Toxicity Criteria (NCI-CTC) version 3.0. Every 2 months, the patients will be evaluated for the clinical effects. If disease progressed, the patients would be ruled out.
  Treatment continued until disease progression, unacceptable toxic effects, patient or physician request to discontinue, or serious protocol non-compliance. A maximum of 2 dose reductions for grade >= 3 toxicity were allowed (100 and 50 mg). A maximum of 2 weeks was permitted for treatment delays due to toxicity.
  Other Names: immunohistochemistry staining method
  Arms: bicalutamide
Other: Physician's Choice — The comparator group, treatment of physician's choice (TPC), represented a mix of agents (both approved and non-approved for metastatic breast cancer) to mirror clinical practice at the time in this setting.
  The 60 patients are enrolled in the study, before randomized to the two arms, each of them will be assessed for eligibility and then their proposed TPC.
  Treatment continued until disease progression, unacceptable toxic effects, patient or physician request to discontinue, or serious protocol non-compliance.
  Arms: Physician's Choice

SUMMARY:
Growing studies demonstrated that Androgen Receptor (AR) has an oncogenic role for the patients with AR-positive Triple Negative Breast Cancer (TNBC). AR antagonists in therapy, such as bicalutamide, completely binds to the AR, increasing AR degradation, thus are investigated for the efficacy of the treatment of patients with AR-positive TNBC in the study.

DETAILED DESCRIPTION:
More than 70% of human breast cancers express the androgen receptor (AR), and in retrospective analysis, the expression of AR in Triple-Negative Breast Cancer (TNBC) varies from 10-43%. Recently emerging preclinical and clinical data suggest that AR may play a role in tumor proliferation. For example, Hu et al (2011) analyzed AR expression in 211 TNBC cases. He found that AR is related with an 83% increase in overall mortality, when compared with AR-negative TNBC. McGhan et al (2014) also found that AR expression tends to exist in TNBC patients with higher tumor stage and lymph metastases.

The role of AR has also been extensively studied in vitro. With targeting AR with small interfering RNA (siRNA) and treatment with anti-androgen bicalutamide, studies showed that AR has a proliferative role in TNBC cells. Robinson et al (2011) also clarified that AR can mimic estrogen receptor α (ERα) in a transcriptionally active manner directed by the forkhead box protein A1 (FoxA1). These indicate that, in ER-negative disease, AR can promote tumor progression, therefore, could serve as a therapeutic target in TNBC.

Due to the demonstration of oncogenic role for the AR in TNBC, clinical trials are underway to study the role of inhibiting androgen signaling for the treatment for TNBC. For example, Gucalp et al (2013) performed a sing-arm phase II study to investigate the role of bicalutamide in AR-positive TNBC. A total of 26 patients were enrolled in the study, and the study demonstrated a general well tolerated effect and a 6-month clinical benefit rate of 19%. Furthermore, future clinical trials are also designed to show the anti-androgen therapy such as Enzalutamide, the 17alpha-hydroxylase/C(17,20)-lyase inhibitor abiraterone acetate and orteronel for AR-positive TNBC. This study is investigated to study the role of bicalutamide for AR-positive TNBC, and it may help clarify the effect of bicalutamide for the specific breast cancer subtype. Furthermore, it may provide an additional therapy to treat the difficult to treat population.

ELIGIBILITY:
Inclusion Criteria:

* Female patients with histologically or cytologically confirmed carcinoma of the breast. Every effort should be made to make paraffin embedded tissue or slides from the diagnostic biopsy or surgical specimen available for confirmation of diagnosis.
* Receptor status: Estrogen receptor- and progesterone receptor-negative,HER-2-negative, Androgen receptor-positive* NOTE: Samples are considered positive if greater than 10% of cell nuclei are immunoreactive.
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 to 2. Life expectancy of >= 3 months.
* Adequate organ and marrow function as defined below:

leukocytes >3,000/mL; absolute neutrophil count >1,500/ml; platelets >100,000/mL; total bilirubin within normal institutional limits; aspartate aminotransferase (AST)/ alanine aminotransferase (ALT) <2.5×institutional upper limit of normal (ULN); creatinine within normal institutional limits OR creatinine clearance >60 mL/min/1.73 m2 for patients with creatinine levels above institutional normal.

* Patients with metastatic disease progressed after one therapeutic regimen for metastatic disease, and there is no limit for the regimens of prior therapy.
* Measurable disease by Response Evaluation Criteria in Solid Tumors (RECIST) criteria.
* Women of childbearing potential, but using (1) surgically sterile or (2) adequate measures of contraception in the opinion of the Investigator. Peri-menopausal women must be amenorrheic for at least 12 months to be considered of non-childbearing potential.
* Patients have no other malignancy, except breast cancer.
* Patients willing and able to comply with the study protocol for the duration of the study.
* Written informed consent prior to any study-specific screening procedures with the understanding that the patient may withdraw consent at any time without prejudice.

Exclusion Criteria:

* Patients who have received any of the following treatments within four weeks before Bicalutamide or TPC treatment start: chemotherapy, radiation, trastuzumab, hormonal therapy, surgery, or any investigational drug within four weeks.
* Patients with a hypersensitivity to Bicalutamide or selected TPC treatment.
* Women who are pregnant or breast-feeding; women of childbearing potential refuse to use any measures of contraception.
* Patients have active brain metastases or leptomeningeal disease.
* Patients have important organ failure or serious marrow suppression.
* Severe/uncontrolled intercurrent illness/infection.
* Significant cardiovascular impairment (history of congestive heart failure > New York Heart Association grade II, severe valvular heart disease，unstable angina or myocardial infarction within the past six months, or serious cardiac arrhythmia, or resistant hypertension).
* Patients can't comply with the study protocol for the duration of the study.
* Patients have had a prior malignancy within five years, other than previous breast cancer.
* Participation in another clinical trial with any investigational agents within 3 weeks prior to study screening.
* Patients with known Central Nervous System (CNS) disease (primary or secondary) or leptomeningeal disease because of their poor prognosis and because they often develop progressive neurological dysfunction that would confound the evaluation of neurological and other adverse events.
* Gastrointestinal disorders interfering with absorption of the study drug.
* Difficulties with swallowing study capsules/tablets.
* Psychiatric disorders or altered mental status precluding understanding of the informed consent process and/or completion of the necessary studies.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2015-01; Primary Completion 2017-01 (Estimated); Study Completion 2017-05 (Estimated)

PRIMARY OUTCOMES:
Clinical benefit rate(CBR) | 1 Year
  The proportion of stability, partial response and complete response in patients who receive bicalutamide as second-, or third-line therapy for estrogen receptor (ER)/ progesterone receptor (PgR)-negative, human epidermal growth factor receptor (HER-2)-negative and AR-positive Metastatic Breast Cancer
Progression-free survival | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 12 months

SECONDARY OUTCOMES:
Quality of life | 1 Year
  FACT(Functional Assessment of Cancer Therapy) -B :a 36-item compilation, subdivided into four primary QOL (Quality of life) domains and a disease specific domain - additional concerns for breast cancer
Number of adverse events (AE) and serious adverse events (SAE) during the course of the study | 1 Year

REFERENCES:
- [Background] Hu R, Dawood S, Holmes MD, Collins LC, Schnitt SJ, Cole K, Marotti JD, Hankinson SE, Colditz GA, Tamimi RM. Androgen receptor expression and breast cancer survival in postmenopausal women. Clin Cancer Res. 2011 Apr 1;17(7):1867-74. doi: 10.1158/1078-0432.CCR-10-2021. Epub 2011 Feb 15. PMID 21325075
- [Background] Robinson JL, Macarthur S, Ross-Innes CS, Tilley WD, Neal DE, Mills IG, Carroll JS. Androgen receptor driven transcription in molecular apocrine breast cancer is mediated by FoxA1. EMBO J. 2011 Jun 24;30(15):3019-27. doi: 10.1038/emboj.2011.216. PMID 21701558
- [Background] McGhan LJ, McCullough AE, Protheroe CA, Dueck AC, Lee JJ, Nunez-Nateras R, Castle EP, Gray RJ, Wasif N, Goetz MP, Hawse JR, Henry TJ, Barrett MT, Cunliffe HE, Pockaj BA. Androgen receptor-positive triple negative breast cancer: a unique breast cancer subtype. Ann Surg Oncol. 2014 Feb;21(2):361-7. doi: 10.1245/s10434-013-3260-7. Epub 2013 Sep 18. PMID 24046116
- [Background] Fioretti FM, Sita-Lumsden A, Bevan CL, Brooke GN. Revising the role of the androgen receptor in breast cancer. J Mol Endocrinol. 2014 Jun;52(3):R257-65. doi: 10.1530/JME-14-0030. Epub 2014 Apr 16. PMID 24740738
- [Background] Shah PD, Gucalp A, Traina TA. The role of the androgen receptor in triple-negative breast cancer. Womens Health (Lond). 2013 Jul;9(4):351-60. doi: 10.2217/whe.13.33. PMID 23826776
- [Background] Gucalp A, Tolaney S, Isakoff SJ, Ingle JN, Liu MC, Carey LA, Blackwell K, Rugo H, Nabell L, Forero A, Stearns V, Doane AS, Danso M, Moynahan ME, Momen LF, Gonzalez JM, Akhtar A, Giri DD, Patil S, Feigin KN, Hudis CA, Traina TA; Translational Breast Cancer Research Consortium (TBCRC 011). Phase II trial of bicalutamide in patients with androgen receptor-positive, estrogen receptor-negative metastatic Breast Cancer. Clin Cancer Res. 2013 Oct 1;19(19):5505-12. doi: 10.1158/1078-0432.CCR-12-3327. Epub 2013 Aug 21. PMID 23965901
- [Background] Park S, Koo J, Park HS, Kim JH, Choi SY, Lee JH, Park BW, Lee KS. Expression of androgen receptors in primary breast cancer. Ann Oncol. 2010 Mar;21(3):488-492. doi: 10.1093/annonc/mdp510. Epub 2009 Nov 3. PMID 19887463
- [Background] Lehmann BD, Bauer JA, Chen X, Sanders ME, Chakravarthy AB, Shyr Y, Pietenpol JA. Identification of human triple-negative breast cancer subtypes and preclinical models for selection of targeted therapies. J Clin Invest. 2011 Jul;121(7):2750-67. doi: 10.1172/JCI45014. PMID 21633166